CLINICAL TRIAL: NCT01030458
Title: Newer vs Older Antihypertensive Agents in African Hypertensive Patients Trial
Brief Title: Newer Versus Older Antihypertensive Agents in African Hypertensive Patients (NOAAH) Trial
Acronym: NOAAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University of Kinshasa (Other); Yaounde Central Hospital (Other Government); University of Yaounde (Other); University of Libreville (Unknown); Institute of Cardiology Abidjan (Unknown); University of Ilorin Teaching Hospital (Other); University of Nigeria, Enugu Campus (Other); Hospital Aristide Le Dantec, Dakar, Senegal (Unknown)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, MD, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOAAH version 5.0.2
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-11

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Hypertension; Blacks; Africa; Blood pressure control; Side-effects
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Valsartan; Amlodipine, Valsartan Drug Combination; Hydrochlorothiazide; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amlodipine plus valsartan (Experimental): In the experimental group, Exforge will be used in two dosage steps, respectively, amlodipine 5 mg plus 160 mg valsartan and amlodipine 10 mg plus 160 mg valsartan.
  Interventions: Drug: amlodipine 5/10 mg per day plus valsartan 160 mg/day
- hydrochlorothiazide plus bisoprolol (Active Comparator): In the reference group, the Lodoz will be used in two dosage steps, respectively 6.25 mg hydrochlorothiazide plus 5 mg or 6.25 mg hydrochlorothiazide plus 10 mg bisoprolol
  Interventions: Drug: hydrochlorothiazide 6.25 mg/day plus bisoprolol 5/10 mg/day

INTERVENTIONS:
Drug: amlodipine 5/10 mg per day plus valsartan 160 mg/day — Amlodipine 5/10 mg/day plus valsartan 160 mg/day, once daily, in the morning
  Other Names: ExForge®
  Arms: amlodipine plus valsartan
Drug: hydrochlorothiazide 6.25 mg/day plus bisoprolol 5/10 mg/day — hydrochlorothiazide 6.25 mg/day plus bisoprolol 5/10 mg/day, once daily, in the morning
  Other Names: Lodoz®
  Arms: hydrochlorothiazide plus bisoprolol

SUMMARY:
The purpose of this study is to compare the blood pressure lowering efficacy of a treatment regimen based on a dihydropyridine calcium-channel blocker combined with an angiotensin II type-1 receptor blocker with the recommended treatment regimen based on a low-dose thiazide diuretic combined with a beta-blocker.

DETAILED DESCRIPTION:
Primary objective:

Sitting systolic blood pressure (average of three readings) will be the primary outcome variable.

Secondary

1. To compare the time interval between the two treatment groups, which after randomisation will be required, to reach and maintain the target defined as a blood pressure below 140 mm Hg systolic and 90 mm Hg diastolic;
2. To compare the duration of follow-up, during which a steady blood pressure control will be achieved;
3. To evaluate the incidence of adverse events, symptoms, biochemical abnormalities and ECG changes in the two treatment groups;
4. To assess the adherence to antihypertensive treatment as well as the rate of drop-outs in both treatment arms during a six-month period.

ELIGIBILITY:
Inclusion Criteria:

* Women or men within an age range from 30 to 69 years with uncomplicated hypertension.
* Blood pressure measured in the sitting position after at least 5 minutes rest (average of three readings at the last run-in-visit) should range from 140 to 179 mm Hg systolic or from 90 to 109 mm Hg diastolic (grades 1 or 2 of hypertension). Patients must have uncomplicated hypertension with a maximum of two additional risk factors, as defined in the 2007 guidelines of the European Societies of Hypertension and Cardiology.
* Systolic blood pressure in the upright position must be at least 110 mm Hg (mean of three readings obtained immediately after the patient has assumed a standing position).
* Patients who have never been treated for hypertension or in whom previous antihypertensive drug treatment has been discontinued for at least four weeks before the last run-in visit can be randomised. If two weeks after discontinuation of previous antihypertensive treatment the blood pressure is higher than 160 mm Hg systolic or higher than 100 mm Hg diastolic and if the patient has complaints, the patient can be randomised immediately to active blood pressure lowering treatment with either the newer or older antihypertensive drugs.
* The patient must provide informed written consent.

Exclusion Criteria:

* Premenopausal women not applying anticonception.
* A history of cardiovascular disease.
* Secondary hypertension.
* Electrocardiographic left ventricular hypertrophy.
* More than two cardiovascular risk factors in addition to hypertension.
* Diabetes mellitus.
* Renal dysfunction.
* Recent treatment with two or more antihypertensive drugs or a contra-indication to discontinue blood pressure lowering agents for 4 weeks.
* Severe non-cardiovascular disease.
* Known contra indications for the first-line study medications.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Kingue, MD, Principal Investigator — Hôpital Général de Yaoundé, BP 5408, Yaoundé, Cameroun; Daniel Lemogoum, MD, PhD, Principal Investigator — Université de Douala, Douala, Cameroon; Bruno Mipinda, MD, Principal Investigator — Hôpital Central Universitaire de Libreville, Libreville, Gabon; Omotoso Babatunde, MD, Principal Investigator — University of Ilorin, Ilorin, Nigeria; Ifeoma E Ulasi, MD, Principal Investigator — University of Enugu, Enugu, Nigeria; Serigne Abdou Ba, MD, Principal Investigator — Hôpital Aristide Le Dantec, Dakar, Sénégal; Jean-René M'Buyamba-Kabangu, MD, PhD, Study Chair — University of Kinshasa, Kinshasa, Democratic Republic of Congo; Jan A Staessen, MD, PhD, Study Director — University of Leuven, Leuven, Belgium
Locations (7):
- Cameroon (2):
  - Ecole de Médecine de Douala, Douala
  - Hôpital Général de Yaoundé, Yaoundé
- Institut de Cardiologie d'Abidjan, Abidjan, Côte d’Ivoire
- Hôpital Central Universitaire de Libreville, Libreville, Gabon
- Nigeria (2):
  - University of Enugu, Enugu
  - University of Ilorin, Ilorin
- Hôpital Aristide Le Dantec, Dakar, Senegal

REFERENCES:
- [Background] Odili AN, Richart T, Thijs L, Kingue S, Boombhi HJ, Lemogoum D, Kaptue J, Kamdem MK, Mipinda JB, Omotoso BA, Kolo PM, Aderibigbe A, Ulasi II, Anisiuba BC, Ijoma CK, Ba SA, Ndiaye MB, Staessen JA, M'buyamba-Kabangu JR; NOAAH Investigators. Rationale and design of the Newer Versus Older Antihypertensive Agents in African Hypertensive Patients (NOAAH) trial. Blood Press. 2011 Oct;20(5):256-66. doi: 10.3109/08037051.2011.572614. Epub 2011 Apr 15. PMID 21495829
- [Result] M'Buyamba-Kabangu JR, Anisiuba BC, Ndiaye MB, Lemogoum D, Jacobs L, Ijoma CK, Thijs L, Boombhi HJ, Kaptue J, Kolo PM, Mipinda JB, Osakwe CE, Odili A, Ezeala-Adikaibe B, Kingue S, Omotoso BA, Ba SA, Ulasi II, Staessen JA; Newer versus Older Antihypertensive Agents in African Hypertensive Patients Trial (NOAAH) Investigators. Efficacy of newer versus older antihypertensive drugs in black patients living in sub-Saharan Africa. J Hum Hypertens. 2013 Dec;27(12):729-35. doi: 10.1038/jhh.2013.56. Epub 2013 Jun 27. PMID 23803591
- [Derived] Osakwe CE, Jacobs L, Anisiuba BC, Ndiaye MB, Lemogoum D, Ijoma CK, Kamdem MM, Thijs L, Boombhi HJ, Kaptue J, Kolo PM, Mipinda JB, Odili AN, Ezeala-Adikaibe B, Kingue S, Omotoso BA, Ba SA, Ulasi II, M'buyamba-Kabangu JR, Staessen JA; Newer Versus Older Antihypertensive Agents in African Hypertensive Patients Trial (NOAAH) Investigators. Heart rate variability on antihypertensive drugs in black patients living in sub-Saharan Africa. Blood Press. 2014 Jun;23(3):174-80. doi: 10.3109/08037051.2013.836810. Epub 2013 Sep 25. PMID 24066715
- [Derived] Odili AN, Ezeala-Adikaibe B, Ndiaye MB, Anisiuba BC, Kamdem MM, Ijoma CK, Kaptue J, Boombhi HJ, Kolo PM, Shu EN, Thijs L, Staessen JA, Omotoso BA, Kingue S, Ba SA, Lemogoum D, M'Buyamba-Kabangu JR, Ulasi II. Progress report on the first sub-Saharan Africa trial of newer versus older antihypertensive drugs in native black patients. Trials. 2012 May 17;13:59. doi: 10.1186/1745-6215-13-59. PMID 22594907

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlodipine Plus Valsartan: In the experimental group, Exforge will be used in two dosage steps, respectively, amlodipine 5 mg plus 160 mg valsartan and to achieve blood pressure control, the study medication could be up-titrated to amlodipine 10 mg plus 160 mg valsartan. Patients take the study medication once a day, in the morning. Follow-up visits will take place at 2 weeks, 1 month and every month thereafter, up until 6 months.
- Hydrochlorothiazide Plus Bisoprolol: In the reference group, the Lodoz will be used in two dosage steps, respectively 6.25 mg hydrochlorothiazide plus 5 mg and to achieve blood pressure control, the study medication could be up-titrated to 6.25 mg hydrochlorothiazide plus 10 mg bisoprolol. Patients take the study medication once a day, in the morning. Follow-up visits will take place at 2 weeks, 1 month and every month thereafter, up until 6 months.
Period: Overall Study
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol
Started | 94 | 89
Completed | 67 | 57
Not Completed | 27 | 32
Not completed — Lost to Follow-up | 9 | 10
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Logistical reasons | 9 | 5
Not completed — Moved or changed job | 6 | 13
Not completed — Side effect of medication | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol | Total
Number analyzed (Participants) | 94 | 89 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 82 | 171
  >=65 years | 5 | 7 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (9.3) | 51.2 (8.7) | 51.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 43 | 96
  Male | 41 | 46 | 87
Region of Enrollment [Number; unit: participants]
  Nigeria | 46 | 46 | 92
  Senegal | 20 | 20 | 40
  Gabon | 6 | 2 | 8
  Cameroon | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Sitting Systolic Blood Pressure on Automated Measurement
Description: Blood pressure is measured by means of validated oscillometric OMRON 705IT recorders (OMRON Healthcare Europe BV, Nieuwegein, Netherlands), after the patient has been seated for 5 minutes in a quiet room, according to the ESC/ESH guidelines. Three consecutive blood pressure readings are obtained and the average of these 3 measurements is used as the primary outcome.
Time Frame: 6 months follow-up after randomization
Population: The main analysis included all randomised patients with at least one follow-up visit, according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol
Number analyzed (Participants) | 94 | 89
mmHg | 127.2 (10.7) | 134.1 (13.1)

2. Secondary Outcome: Time to Blood Pressure Control
Description: The time (in weeks) after randomisation that will be required to reach and maintain the target, defined as a blood pressure below 140 mmHg systolic and 90 mmHg diastolic.
Time Frame: 6 months follow-up after randomization
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol
Number analyzed (Participants) | 94 | 89
weeks | 12 [4 to 20] | 18 [4 to 24]

3. Secondary Outcome: Side-effects to Study Medications
Time Frame: 6 months follow-up after randomization
Measure: Number; unit: participants
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol
Number analyzed (Participants) | 94 | 89
participants | 1 | 1

4. Secondary Outcome: Proportion of Patients Reaching Blood Pressure Control at the End of Follow-up
Description: This variable gives the proportion of patients reaching blood pressure control over time (< 140 mmHg systolic and < 90 mmHg diastolic)
Time Frame: 6 months follow-up after randomization
Measure: Number; unit: participants
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol
Number analyzed (Participants) | 94 | 89
participants | 58 [4 to 20] | 40 [4 to 24]

ADVERSE EVENTS:
Arm/Group | Amlodipine Plus Valsartan | Hydrochlorothiazide Plus Bisoprolol
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/89
Other Adverse Events (participants affected / at risk) | 1/94 | 1/89
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine Plus Valsartan (N=94) | Hydrochlorothiazide Plus Bisoprolol (N=89)
Insomnia/asthenia (Nervous system disorders) | 0 (0) | 1 (1)
Bilateral leg oedema (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No